CLINICAL TRIAL: NCT04251039
Title: "Efficacy and Safety of Oral/iv Therapy (Cangrelor) in Patients With SCAD Undergoing Complex PCI, the RESPONSE Study"
Brief Title: in Patients With SCAD Undergoing Complex PCI, the RESPONSE Study"
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fondazione GISE Onlus (Other)
Responsible Party: Sponsor
Other Study IDs: RESPONSE V 0.4 31/10/2019
Record Dates: First submitted 2020-01-03; First posted 2020-01-31 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- PCI with pre-treatment with P2Y12 inhibitors: SCAD patients undergoing complex PCI with pre-treatment with P2Y12 inhibitors will undergo:
  * Assessment of platelet reactivity (Time 0, T0) (VFN)
  * PCI (start = T1; end= T2)
- PCI with treatment with P2Y12 inhibitors only after procedure.: SCAD patients undergoing complex PCI with treatment with P2Y12 inhibitors only after procedure will undergo:
  * Administration of Cangrelor (bolus + infusion of at least 2 hours and at least until end of PCI) or decision to not administer (T0)
  * Assessment of platelet reactivity (Time 0, T0) (VFN)
  * PCI (start of PCI= T1; end of infusion of Cangrelor= T2)

SUMMARY:
Evaluation of Efficacy/Safety in Cangrelor use in patients with SCAD undergoing complex PCI.

Prospective, observational, multicenter registry.

DETAILED DESCRIPTION:
SCAD patients routinely in the Italian centers undergo complex PCIs with pre-treatment with P2Y12 inhibitors or with P2Y12 inhibitors administration after procedure. This implies that participants receive interventions as part of routine medical care, and that researchers actually observe the effect of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 65 years of age at the time of signing the Informed Consent Form
* Patient presenting with SCAD undergoing complex PCI and:

  * Type 2 Diabetes Mellitus;
  * CKD (Grade specified in CRF);
  * Complex SCAD: LMD, 3VD, bifurcation lesions, Rotablator, CTO, multiple Stents, total length of the stents must be greater than 60 mm.
* Patient is to be treated for de novo lesions located in previously untreated vessels.
* Patient must agree to undergo all required follow-up visits and data collection.

Exclusion Criteria:

* History of CABG;
* In stent restenosis;
* Patient with intolerance or contra-indications to treatment with aspirin, clopidogrel, prasugrel, ticagrelor, cangrelor, heparin, contrast media;
* Patient on chronic treatment with oral anticoagulants;
* Patient with neoplastic or rheumatic diseases;
* Use of dipyridamole, cilostazol, or anticoagulant therapy during the study period;
* Bleeding disorder
* History of an ischemic stroke or intracranial bleeding
* Intracranial vascular abnormality;
* Gastrointestinal bleeding within the previous 6 months or major surgery within the previous 30 days.
* Women who are pregnant/breastfeeding or who have the potential to become pregnant during the study;
* Patient with bleeding diathesis in whom antiplatelet drug is contraindicated;
* Concomitant indication to open heart surgery
* Inability to provide written informed consent
* Enrolment in another study within 1 month

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with SCAD undergoing complex PCI
Sampling Method: Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Safety endpoint: Major bleedings according with Thrombolysis in Myocardial Infarction (TIMI) classification. | hour 48
  Number of patients with intracranial hemorrhage or a ≥5 g/dl decrease in hemoglobin concentration or a ≥15 % absolute decrease in hematocrit.

SECONDARY OUTCOMES:
Efficacy endpoint: Long-term major adverse cardiac and cerebrovascular events MACCE (eg Death from any cause, Any Myocardial infarction, Revascularization, Stroke) | hour 48 and day 30
  Number of patients with Long-term major adverse cardiac and cerebrovascular events (MACCE) (e.g. Death from any cause, Any Myocardial infarction, Revascularization, Stroke)
Assessment of platelet reactivity | Day 0
  Assessment of platelet reactivity measured by the VerifyNow® P2Y12 assay. Pharmacodynamic measurements will occur according to manufacturer instructions before, during, and after study drug infusion.
Number of Participants with stent thrombosis | hour 48
  Number of Participants with stent thrombosis demonstrated by coronary angiography
Rehospitalisation due to unstable or progressive angina according to the Braunwald Unstable Angina Classification and the Canadian Cardiovascular Society Angina Classification. | Day 30
  Rehospitalisation due to unstable or progressive angina according to the Braunwald Unstable Angina Classification and the Canadian Cardiovascular Society Angina Classification.
Time to Coronary Artery Bypass Graft (CABG) | Day 30
  Time between the intervention and the Coronary Artery Bypass Graft (CABG)

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Marchese, MD, PhD, Principal Investigator — Ospedale Santa Maria (BA)
Locations (1):
- Ospedale Santa Maria, Bari, Apulia, Italy